CLINICAL TRIAL: NCT05008432
Title: Sleep Apnea in Heart Failure With Preserved Ejection Fraction - Exercise Capacity and Impact of Positive Airway Pressure Therapy
Brief Title: Sleep Apnea in Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Itamar-Medical, Israel (Industry); Sleep Number Corporation (Unknown)
Responsible Party: Principal Investigator, Yogesh Reddy, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 21-002139
Record Dates: First submitted 2021-07-15; First posted 2021-08-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Obstructive Sleep Apnea
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFpEF Patients Diagnosed with Obstructive Sleep Apnea: Right heart cath patients who are diagnosed with HFpEF will undergo a home sleep apnea test (for patients hospitalized with HFpEF, the initial home sleep test will be performed in hospital overnight)
  Interventions: Diagnostic Test: Home sleep apnea testing

INTERVENTIONS:
Diagnostic Test: Home sleep apnea testing — Participants will be monitored with a WatchPAT device for home based diagnosis of OSA (for patients hospitalized with HFpEF, the sleep test may be performed in the hospital or at home).

SUMMARY:
This is a prospective interventional study to better understand i) the prevalence of Obstructive Sleep Apnea (OSA) in Heart Failure with preserved Ejection Fraction (HFpEF), ii) its hemodynamic correlates, and iii) the impact of intervention with Continuous Positive Airway Pressure (CPAP) on quality of life.

DETAILED DESCRIPTION:
This is a prospective non-randomized observational study which will recruit patients with gold standard HFpEF defined by exercise catheterization or following HF hospitalization. The prevalence of OSA will be determined in all HFpEF patients at baseline using home sleep apnea testing and all patients will complete the Mayo Sleep Questionnaire. Patients with known OSA at baseline will also be included only for the baseline assessment to accurately estimate prevalence of OSA in gold standard diagnosed HFpEF. The subset of initially recruited patients with HFpEF who have newly diagnosed OSA will be offered and initiated on CPAP therapy to treat their underlying OSA. Repeat evaluation after 3 months of CPAP therapy for end point assessment with remote accelerometry (2 weeks prior to study completion), ESS and KCCQ, which will all be identical to baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of HFpEF by catheterization with resting PCWP>15 mmHg or exercise PCWP>25 mmHg or hospitalization with HFpEF
* Ambulatory (not wheelchair/scooter dependent)
* If no known diagnosis of OSA, must not be pacemaker dependent with either atrial pacing or VVI without sinus rhythm
* If no known diagnosis of OSA, must be able to temporarily hold nitrates or alpha channel blockers for home WatchPAT testing (3 hour washout period)

Exclusion Criteria:

* Ejection fraction <40%
* Obstructive hypertrophic cardiomyopathy
* Constrictive pericarditis or tamponade
* Active myocarditis
* Complex congenital heart disease
* Other valve disease requiring surgical intervention
* Terminal illness (other than HF) with expected survival of less than 1 year
* Inability to comply with planned study procedures
* Pregnancy or breastfeeding mothers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Determine the impact of intervention with CPAP therapy on quality of life as assessed by Kansas City Cardiomyopathy Questionnaire scores (Scale 0-100) in patients with Obstructive Sleep Apnea at Baseline | 6 months
  Quality of life will be assessed by Kansas City Cardiomyopathy Questionnaire (Scale 0-100)

SECONDARY OUTCOMES:
Determine the impact of intervention with CPAP therapy on average daily accelerometry units (scale -1000 to 10000 units) by wearable accelerometers in patients with Obstructive Sleep Apnea at Baseline | 6 months
  Average daily accelerometry units by wearable accelerometers (scale -1000 to 10000 units)
Determine the impact of intervention with CPAP therapy on hours active per day (number of hours of activity per day range 0-12 hours) by wearable accelerometers in patients with Obstructive Sleep Apnea at Baseline | 6 months
  Hours of activity per day by wearable accelerometers (number of hours of activity per day range 0-12 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Reddy, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials